CLINICAL TRIAL: NCT06202534
Title: An Observational Clinical Study Plan on the Effects of Radiotherapy on the Immune System of Patients With Malignant Tumors.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Yong Wu, An Observational Clinical Study Plan on the Effects of Radiotherapy on the Immune System of Patients With Malignant Tumors., Guangzhou First People's Hospital
Other Study IDs: K-2023-093-01
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Malignant Neoplasm
Keywords: Erythroid Precursor Cells
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Before radiotherapy,: Samples were collected from patients with breast cancer, nasopharyngeal cancer, colorectal cancer, cervical cancer, lung cancer, and head and neck cancer. 5 ml of peripheral blood was extracted from these patients before radiotherapy, and flow cytometry was used to detect MDSCs, T cells, and erythroid precursor cells.
- During radiotherapy: Samples were collected from patients with breast cancer, nasopharyngeal cancer, colorectal cancer, cervical cancer, lung cancer, and head and neck cancer. 5 ml of peripheral blood was extracted from these patients during radiotherapy, and flow cytometry was used to detect MDSCs, T cells, and erythroid precursor cells.
- After radiotherapy: Samples were collected from patients with breast cancer, nasopharyngeal cancer, colorectal cancer, cervical cancer, lung cancer, and head and neck cancer. 5 ml of peripheral blood was extracted from these patients after radiotherapy, and flow cytometry was used to detect MDSCs, T cells, and erythroid precursor cells.
- 3 months after radiotherapy: Samples were collected from patients with breast cancer, nasopharyngeal cancer, colorectal cancer, cervical cancer, lung cancer, and head and neck cancer. 5 ml of peripheral blood was extracted from these patients 3 months after radiotherapy, and flow cytometry was used to detect MDSCs, T cells, and erythroid precursor cells.

INTERVENTIONS:
Other:  — radiotherapy

SUMMARY:
To explore the impact of radiotherapy on peripheral blood myeloid-derived suppressor cells (MDSCs), T cells and extramedullary erythroid precursor cells in patients with malignant tumors, and to evaluate the correlation between changes in the proportion of these cells before and after radiotherapy and the efficacy of radiotherapy in patients.

DETAILED DESCRIPTION:
To clarify the impact of radiotherapy (and/or other treatment combinations) on the proportion of myeloid-derived suppressor cells (MDSCs), T cells and extramedullary erythroid precursor cells in the peripheral blood of patients with malignant tumors, and to evaluate the changes in the proportion of these cells before and after radiotherapy and the relationship between the patients Correlation with the efficacy of radiotherapy. On this basis, it provides theoretical guidance for the determination of new clinical treatment plans.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old, diagnosed with breast cancer, nasopharyngeal cancer, colorectal cancer, cervical cancer, lung cancer, head and neck cancer and requiring radiotherapy, and the above malignant tumors have not metastasized.
2. Complete inspection information.
3. No other serious complications.
4. No infectious diseases.
5. Able and willing to take blood tests.
6. All researchers gave informed consent and signed an informed consent form, which complied with the requirements of the Medical Ethics Committee.

Exclusion Criteria:

1. People with mental illness.
2. People with autoimmune system diseases.
3. Those combined with serious diseases of other organs.
4. Those with severe alcoholism and drug abuse.
5. Research subjects who voluntarily withdraw from the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Over 18 years old, diagnosed with breast cancer, nasopharyngeal cancer, colorectal cancer, cervical cancer, lung cancer, head and neck cancer and requiring radiotherapy, and the above malignant tumors have not metastasized.
  2. Complete inspection information.
  3. No other serious complications.
  4. No infectious diseases.
  5. Able and willing to take blood tests.
  6. All researchers gave informed consent and signed an informed consent form, which complied with the requirements of the Medical Ethics Committee.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Erythroid precursor cells increase after radiotherapy. | Erythroid precursor cells increase after radiotherapy.Erythroid precursor cells gradually decreased to the pre-radiation level after 3 months of radiotherapy.
  Erythroid precursor cells increase after radiotherapy.Erythroid precursor cells gradually decreased to the pre-radiation level after 3 months of radiotherapy.

SECONDARY OUTCOMES:
Peripheral blood myeloid-derived suppressor cells (MDSCs) increase after radiotherapy. | Peripheral blood myeloid-derived suppressor cells (MDSCs) increase after radiotherapy.Peripheral blood myeloid-derived suppressor cells (MDSCs) gradually decreased to the pre-radiation level after 3 months of radiotherapy.
  Peripheral blood myeloid-derived suppressor cells (MDSCs) increase after radiotherapy.Peripheral blood myeloid-derived suppressor cells (MDSCs) gradually decreased to the pre-radiation level after 3 months of radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- GuangzhouFPH, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No